CLINICAL TRIAL: NCT00077233
Title: A Phase II Trial Of Irinotecan /5-FU/ Leucovorin Or Oxaliplatin /5-FU / Leucovorin With And Without Cetuximab (C225) For Patients With Untreated Metastatic Adenocarcinoma Of The Colon or Rectum
Brief Title: FOLFIRI or FOLFOX With or Without Cetuximab in Patients With Metastatic Adenocarcinoma of the Colon or Rectum
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Bristol-Myers Squibb (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB 80203; U10CA031946 (NIH); CDR0000350016 (Other: Physician Data Query)
Record Dates: First submitted 2004-02-10; First posted 2004-02-11 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the colon; adenocarcinoma of the rectum; recurrent colon cancer; recurrent rectal cancer; stage IV colon cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Cetuximab; Fluorouracil; Irinotecan; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm A: FOLFIRI (Active Comparator): Patients receive irinotecan 180 mg/m^2 over 90 minutes on day 1, then leucovorin 400 mg/m^2 over 2 hours followed by 5FU 400 mg/m^2 IV bolus injection then 5FU 2400 mg/m^2 continuous IV infusion over 46-48 hours repeated every 2 weeks. One cycle of therapy is 8 weeks.
  Interventions: Drug: 5-FU; Drug: irinotecan; Drug: leucovorin
- Arm B: FOLFIRI + C225 (Experimental): Patients receive irinotecan 180 mg/m^2 over 90 minutes, then leucovorin 400 mg/m^2 IV over 2 hours followed by 5FU 400 mg/m^2 IV bolus injection then 5FU 2400 mg/m^2 continuous IV infusion over 46-48 hours repeated every 2 weeks. Patients also receive cetuximab 400 mg/m^2 IV over 120 minutes day 1, then 250 mg/m^2 IV over 60 minutes weekly. All patients must be premedicated with diphenhydramine hydrochloride 50 mg (or a similar agent) IV prior to the first dose of cetuximab in an effort to prevent a hypersensitivity reaction. Premedication is recommended prior to subsequent doses, but at the Investigator's discretion the dose of diphenhydramine (or a similar agent) may be reduced.
  Interventions: Drug: cetuximab; Drug: 5-FU; Drug: irinotecan; Drug: leucovorin
- Arm C: FOLFOX (Active Comparator): Patients receive oxaliplatin 85 mg/m^2 IV infused over 120 minutes, then leucovorin 400 mg/m^2 IV over 2 hours followed by 5 FU 400 mg/m^2 IV bolus injection then 5 FU 2400 mg/m^2 continuous IV infusion over 46-48 hours every 2 weeks.
  Interventions: Drug: 5-FU; Drug: leucovorin; Drug: oxaliplatin
- Arm D: FOLFOX + C225 (Experimental): Patients receive oxaliplatin 85 mg/m^2 IV infused over 120 minutes, then leucovorin 400 mg/m^2 over 2 hours followed by 5 FU 400 mg/m^2 IV bolus injection then 5 FU 2400 mg/m^2 continuous IV infusion over 46-48 hours every 2 weeks. Patients also receive cetuximab 400 mg/m^2 IV over 120 minutes day 1, then 250 mg/m^2 IV over 60 minutes weekly. All patients must be premedicated with diphenhydramine hydrochloride 50 mg (or a similar agent) IV prior to the first dose of cetuximab in an effort to prevent a hypersensitivity reaction. Premedication is recommended prior to subsequent doses, but at the Investigator's discretion the dose of diphenhydramine (or a similar agent) may be reduced.
  Interventions: Drug: cetuximab; Drug: 5-FU; Drug: leucovorin; Drug: oxaliplatin

INTERVENTIONS:
Drug: cetuximab — IV
  Other Names: C225
  Arms: Arm B: FOLFIRI + C225; Arm D: FOLFOX + C225
Drug: 5-FU — IV
  Other Names: 5-fluorouracil
Drug: irinotecan — IV
  Other Names: CPT-11
  Arms: Arm A: FOLFIRI; Arm B: FOLFIRI + C225
Drug: leucovorin — IV
  Other Names: calcium folinate
Drug: oxaliplatin — IV
  Other Names: Eloxatin
  Arms: Arm C: FOLFOX; Arm D: FOLFOX + C225

SUMMARY:
This is a randomized phase II study trial that has served as a screening trial to test the increased efficacy of chemotherapy + cetuximab versus chemotherapy alone among patients with untreated, advanced or metastatic colon cancer regardless of tumor status with respect to EGFR.

DETAILED DESCRIPTION:
CALGB 80203 was activated on December 15, 2003. In February 2004, based on the results of the randomized trial of IFL +/- cetuximab showing a significant improvement in overall survival with cetuximab, cetuximab was approved by the FDA for use as front-line therapy for patients with metastatic colon cancer. In response to this action, the Data Safety and Monitoring Board recommended closure of CALGB 80203. CALGB 80203 was subsequently closed to accrual in January 2005 with 238 of the originally targeted 2200 patients enrolled. A final decision was to "replace" CALGB 80203 with a three-treatment arm randomized trial of chemotherapy (FOLFOX or FOLFIRI) with and without cetuximab and/or bevacizumab. The protocol was amended to allow analysis of the data from CALGB 80203 as a randomized phase II trial and reporting of the results.

Patients were stratified according to prior adjuvant chemotherapy (yes vs no) and prior pelvic radiation (yes vs no). Patients must have completed any major surgery or radiotherapy (eg, chest or bone palliative RT or pelvic RT) ≥ 4 weeks from registration and completed any minor surgery ≥ 2 weeks from registration. Patients must have fully recovered from the procedure and/or radiotherapy. Patients must have initiated treatment within 7 days of registration. Patients were randomized to 1 of 4 treatment arms, please see a description of the treatment regimens in the "Arms" section. In addition, patients received concomitant and supportive therapy as appropriate per the protocol.

OBJECTIVES:

Primary

1. To determine if the addition of C225 to FOLFIRI or FOLFOX chemotherapy prolongs survival of patients with untreated, advanced or metastatic colorectal cancer.

Secondary

1. To determine if the FOLFIRI and FOLFOX regimens are equivalent in terms of survival as front-line therapy for advanced colorectal patients.
2. To determine the level of EGFR expression in patients with metastatic colorectal cancer.

Patients were followed up to 3 years post-treatment.

ELIGIBILITY:
1. Locally Advanced or Metastatic Colorectal Cancer

   * Eligible patients must have histologically or cytologically documented locally advanced or metastatic colorectal cancer. The site of the primary lesion must be or have been confirmed endoscopically, surgically or radiologically to have been in the large bowel.
   * Patients with a history of colorectal cancer treatment by surgical resection who develop radiological or clinical evidence of metastatic cancer do not require separate histological or cytological confirmation of metastatic disease unless:

     * Either an interval of greater than five years has elapsed between the primary surgery and the development of metastatic disease OR
     * The primary cancer was stage I.
   * Clinicians should consider biopsy of lesions to establish the diagnosis of metastatic colorectal cancer in each case if there is substantial clinical ambiguity regarding the nature or source of apparent metastases.
2. No prior treatment for advanced or metastatic colorectal cancer

   * Patients may have received prior adjuvant chemotherapy (no more than 6 months or 4 cycles) or radiation with radiosensitizing chemotherapy. The last course of chemotherapy must have concluded > 12 months prior to registration. Patients may not have previously received irinotecan ≤ or oxaliplatin therapy in either the adjuvant or metastatic setting. No concurrent use of additional investigational agents is allowed while participating in this study.
3. Patients may not have had prior radiotherapy to greater than 25% of bone marrow.

   Standard adjuvant rectal cancer chemoradiation will not exclude the patient from protocol entry. Radiation must have concluded ≥ 4 weeks from registration.
4. Patients should have completed any major surgery ≥ 4 weeks from registration. Patients must have completed any minor surgery ≥ 2 weeks from registration. Patients must have fully recovered from the procedure. Insertion of a vascular access device is not considered major or minor surgery.
5. No previous or concurrent malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for five years.
6. Age ≥ 18 years
7. CTC (ECOG) performance status of 0-1.
8. No evidence of Gilbert's syndrome - Patients with Gilbert's Syndrome may have a greater risk of irinotecan toxicity due to the abnormal glucuronidation of SN-38. Evidence of Gilbert's Syndrome would include a prior finding of an isolated elevation of indirect bilirubin.
9. Patients must have at least one paraffin block available or appropriate number of unstained slides for analysis of EGFR status.
10. No symptomatic sensory peripheral neuropathy of ≥ grade II at baseline.
11. Non-pregnant and non-lactating

    * Women of child bearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG within 72 hours prior to initiation of treatment. This is because DNA alkylating agents are known to be teratogenic, and the effects of irinotecan, OXAL, 5-FU and C225 on a developing fetus at the recommended therapeutic doses are unknown.
    * Women of child bearing potential includes:

      * any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or
      * is not postmenopausal [defined as amenorrhea ≥ 12 consecutive months] or
      * women on hormone replacement therapy [HRT] with documented serum follicle stimulating hormone (FSH) level > 35 mIU/mL
      * women who are using oral, implanted or injectable contraceptive hormones or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy or practicing abstinence or where partner is sterile (eg, vasectomy), should be considered to be of child bearing potential.
    * Should a woman become pregnant or suspect she is pregnant while participating on on this study, she should inform her physician immediately. Because the risk of toxicity of these agents in nursing infants is also unknown, breastfeeding should be discontinued.
12. No known central nervous system metastases or carcinomatous meningitis.
13. No interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung.
14. No pleural effusion or ascites that causes ≥ grade 2 dyspnea.
15. No predisposing colonic or small bowel disorders in which the symptoms are uncontrolled as indicated by baseline pattern of > 3 watery or soft stools daily in patients without a colostomy or ileostomy. Patients with a colostomy or ileostomy may be entered at investigator discretion.
16. No prior exposure or known sensitivity to chimerized or murine antibodies, C225 (or other EGFR inhibitors) or any tyrosine kinase inhibitors
17. No significant history of cardiac disease, such as unstable angina, CHF, MI, stroke or a LVEF below the institutional range of normal on a baseline multiple gated acquisition (MUGA) or echocardiogram.
18. Patients must not have an uncontrolled seizure disorder, or active neurological disease.
19. Patients may not have received itraconazole or ketoconazole less than 4 weeks prior to registration.
20. Required Initial Laboratory Values:

    * Granulocytes ≥ 1500/ µl
    * Hemoglobin ≥ 9.0 gram/dL (patient may be transfused to meet this criterion)
    * Platelet count ≥ 100,000/ µl
    * Creatinine ≤ 1.5 x Upper limits of normal (ULN)
    * Bilirubin ≤ 1.5 mg/dL
    * AST ≤ 5.0 x ULN
    * Albumin ≥ 2.5 gram/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2003-12; Primary Completion 2006-12 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Overall survival | Up to 3 years of follow up

SECONDARY OUTCOMES:
Progression-free survival | Up to 18 months of follow up
Complete response | Up to 18 months of follow up
Partial response | Up to 18 months of follow up
Proportion of patients experiencing ≥ Grade 3 diarrhea | Up to 30 days post-treatment
Proportion of patients experiencing ≥ Grade 3 ANC | Up to 30 days post-treatment
Percent of total dose administered | Up to 30 days post-treatment
Proportion of patients experiencing ≥ Grade 4 toxicity on each cetuximab treatment arm | Up to 30 days post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Alan Venook, MD, Study Chair — University of California, San Francisco
Locations (77):
- United States (77):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Cedars-Sinai Comprehensive Cancer Center at Cedars-Sinai Medical Center, Los Angeles, California
  - Naval Medical Center - San Diego, San Diego, California
  - Veterans Affairs Medical Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Washington, DC, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Memorial Regional Cancer Center at Memorial Regional Hospital, Hollywood, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Fort Wayne Medical Oncology and Hematology, Incorporated, Fort Wayne, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Baptist Hospital East - Louisville, Louisville, Kentucky
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - Lakeland Cancer Care Center at Lakeland Hospital - St. Joseph, Saint Joseph, Michigan
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - Las Vegas, Las Vegas, Nevada
  - New Hampshire Oncology-Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper University Hospital, Camden, New Jersey
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., East Syracuse, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Veterans Affairs Medical Center - Asheville, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - NorthEast Oncology Associates - Concord, Concord, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - FirstHealth Moore Regional Hospital, Pinehurst, North Carolina
  - Zimmer Cancer Center at New Hanover Regional Medical Center, Wilmington, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital at Ohio State University, Columbus, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Lifespan: The Miriam Hospital, Providence, Rhode Island
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Simmons Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Virginia Oncology Associates - Norfolk, Norfolk, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Incorporated - Roanoke, Roanoke, Virginia
  - St. Mary's Medical Center, Huntington, West Virginia

REFERENCES:
- [Result] Meyerhardt JA, Jackson McCleary N, Niedzwiecki D, et al.: Impact of age and comorbidities on treatment effect, tolerance, and toxicity in metastatic colorectal cancer (mCRC) patients treated on CALGB 80203. [Abstract] J Clin Oncol 27 ( Suppl 15): A-4038, 2009.
- [Result] Venook A, Niedzwiecki D, Hollis D, et al.: Phase III study of irinotecan/5FU/LV (FOLFIRI) or oxaliplatin/5FU/LV (FOLFOX) ± cetuximab for patients (pts) with untreated metastatic adenocarcinoma of the colon or rectum (MCRC): CALGB 80203 preliminary results. [Abstract] J Clin Oncol 24 (Suppl 18): A-3509, 2006.